CLINICAL TRIAL: NCT04348227
Title: How COVID-19 Virus Outbreak Affects Antimicrobial Resistance in a Low-middle-income Country's ICU?
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: Hôpital Universitaire Fattouma Bourguiba (Other)
Responsible Party: Principal Investigator, Khemili Malek, Principal investigator, Hôpital Universitaire Fattouma Bourguiba
Other Study IDs: KM2020-1
Record Dates: First submitted 2020-04-10; First posted 2020-04-16 (Actual); Last update posted 2020-04-17 (Actual); Status verified 2020-04

CONDITIONS: Ventilator Associated Pneumonia
MeSH Terms: conditions — Pneumonia, Ventilator-Associated

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Other
Patient Registry: Yes
Target Follow-Up Duration: 2 Years
Biospecimen Retention: Samples Without DNA — Endotracheal aspirates
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Before pandemic is declared: Positive endotracheal aspirates addressed from January 1st 2019 to January 1st 2020
- After pandemic is declared: Positive endotracheal aspirates addressed from February1st 2020 to February 1st 2021
  Interventions: Behavioral: Enhanced hygiene measures

INTERVENTIONS:
Behavioral: Enhanced hygiene measures — Wether or not hygiene measures dictated by the pandemic of severe acute respiratory syndrome coronavirus 19 , reduce multi drug resistant pathogens isolated in endotracheal aspirates.
  Groups: After pandemic is declared

SUMMARY:
A previous study showed a high incidence of ventilator-associated pneumonia to multidrug resistant pathogens in our ICU. That has been related to lack of compliance to hand hygiene among health care providers in ou ICU.

DETAILED DESCRIPTION:
A single-center cohort study performed in the department of Anesthesia and Intensive Care in our Hospital. All endotracheal isolates realised in the period of study are collected from the Department of Microbiology of our Hospital.

ELIGIBILITY:
Inclusion Criteria:

* Patients requiring mechanical ventilation for more than 24 hours

Exclusion Criteria:

-

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: All patients admitted in ICU in the period of the study, requiring mechanical ventilation for more than 24 hours
Sampling Method: Non-Probability Sample
Enrollment: 120 (Estimated)
Dates: Start 2019-01-01 (Actual); Primary Completion 2020-01-01 (Actual); Study Completion 2021-02-04 (Estimated)

PRIMARY OUTCOMES:
MDR pathogens in endotracheal aspirates | 1 year
  Incidence of MDR bacteria in endotracheal aspirates

SECONDARY OUTCOMES:
Microorganisms in endotracheal aspirates | 1 year
  Incidence of microorganisms in endotracheal aspirates

CONTACTS AND LOCATIONS:
Overall Officials: Malek Khemili, Resident, Principal Investigator — Department of anesthesia and intensive care, Fattouma Bourguiba Hospital
Locations (1):
- Department of anesthesia and intensive care, Fattouma Bourguiba Hospital, Monastir, Tunisia

IPD SHARING:
Plan to Share IPD: Undecided